CLINICAL TRIAL: NCT03268239
Title: Contrast-enhanced 3D T1-weighted Gradient-echo Versus Spin-echo 3 Tesla MR Sequences in the Detection of Active Multiple Sclerosis Lesions
Acronym: COGITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALR_2017_11
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Magnetic Resonance Imaging; Central Nervous System; Brain; Multiple Sclerosis; Demyelinating Diseases
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI sequences (Other): There will be only one arm of patients with central nervous system inflammatory disease.
  Each patient will be its own control. The usual and additional MRI sequences will be performed in all patients and the number of lesions obtained in usual sequences and additional sequences will be compared in the same patient.
  Interventions: Device: Additional MRI sequences

INTERVENTIONS:
Device: Additional MRI sequences — Due to the participation in the study, the following sequences are added to the imaging protocol:
  * 3D T1 GRE after injection (Gradient-Recalled Echo)
  * 3D T1 TSE before injection (Turbo Spin Echo)
  * 3D fGATIR PSIR after injection (fast Gray Matter Acquisition T1 Inversion Recovery Phase-Sensitive Inversion Recovery)
  Sequences will be performed in a random order to avoid the bias induced by different time intervals between injection and acquisition.

SUMMARY:
Gadolinium-enhanced magnetic resonance imaging (MRI) is currently the imaging gold standard to detect active inflammatory lesions in multiple sclerosis (MS) patients. The sensitivity of enhanced MRI to detect active lesions may vary according to the acquisition strategy used (e.g., delay between injection and image acquisition, contrast dose, field strength, and frequency of MRI sampling). Selection of the most appropriate T1-weighted sequence after contrast injection may also influence sensitivity. Several clinical studies performed at 1.5 Tesla have shown that conventional 2D spin-echo (SE) sequences perform better than gradient recalled-echo (GRE) sequences for depicting active MS lesions after gadolinium injection. As relates to MS, 3.0 Tesla systems offer some advantages over lower field strengths, such as higher detection rates for T2 and gadolinium-enhancing brain lesions, an important capability for diagnosing and monitoring MS patients. Recent studies have shown that at 3 Tesla, 3D GRE or 3D fast SE sequences provide higher detection rates for gadolinium-enhancing MS lesions, especially smaller ones, than standard 2D SE, and better suppress artefacts related to vascular pulsation. However, the comparison of the performance of 3D GRE versus 3D SE sequences has not been investigated yet.

Objectives To compare the sensitivity of enhancing multiple sclerosis (MS) lesions in gadolinium-enhanced 3D T1-weighted gradient-echo (GRE) and turbo-spin-echo (TSE) sequences.

ELIGIBILITY:
Inclusion Criteria:

* Equal or more than 18 years of age
* Able to provide written informed consent.
* Known central nervous system inflammatory disease
* Magnetic Resonance exam needed for evaluation after a clinical event in the last 3 weeks

Exclusion Criteria:

* Current treatment with dimethylfumarate (Tecfidera®), natalizumab (Tysabri®) or fingolimod (Gilenya®)
* Contraindications either to 3 Tesla Magnetic Resonance Imaging (e.g. certain metallic and electronic implants, claustrophobia) or IV gadolinium contrast (allergy, pregnancy, breast-feeding, renal insufficiency).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Number of gadolinium-enhanced brain lesions | Baseline
  Number of gadolinium-enhanced brain lesions depicted on a 3D T1 Turbo Spin Echo sequence compared to those depicted on the 3D T1 Gradient-Recalled Echo sequence.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] de Panafieu A, Lecler A, Goujon A, Krystal S, Gueguen A, Sadik JC, Savatovsky J, Duron L. Contrast-Enhanced 3D Spin Echo T1-Weighted Sequence Outperforms 3D Gradient Echo T1-Weighted Sequence for the Detection of Multiple Sclerosis Lesions on 3.0 T Brain MRI. Invest Radiol. 2023 May 1;58(5):314-319. doi: 10.1097/RLI.0000000000000937. Epub 2022 Dec 8. PMID 36729811